CLINICAL TRIAL: NCT00120094
Title: ISSUE 2. The Management of Patients With Suspected or Certain Neurally-Mediated Syncope After the Initial Evaluation
Brief Title: International Study on Syncope of Uncertain Etiology
Status: Terminated | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Medtronic (Industry)
Other Study IDs: ISS2
Record Dates: First submitted 2005-06-30; First posted 2005-07-15 (Estimated); Last update posted 2006-04-11 (Estimated); Status verified 2005-07

CONDITIONS: Syncope
Keywords: Syncope; Electrocardiographic monitoring
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This is a multi-center, prospective, observational study enrolling 400 patients with suspected or certain neurally-mediated syncope, who undergo carotid sinus massage, tilt testing and Implantable Loop Recorder (ILR)implantation. In its second phase, which starts after the first ILR-documented syncope, the study will register the patient outcome after administration of ILR-guided therapy, which is left to the discretion of the physicians. The main objective is to verify the value of ILR in assessing the mechanism of syncope and the efficacy of the ILR-guided therapy after syncope recurrence.

DETAILED DESCRIPTION:
Study purpose was to verify the value of an Implanted Loop Recorder (ILR) in assessing the mechanism of syncope and the efficacy of ILR-guided therapy after documentation of syncope recurrence in patients with suspected or certain neurally-mediated syncope at initial evaluation.

Multi-center, prospective, observational study enrolling 400 patients with suspected or certain neurally-mediated syncope, who undergo carotid sinus massage, tilt testing and ILR implantation. In its second phase, which starts after the first ILR-documented syncope, the study will register the patient outcome after administration of ILR-guided therapy, which is left to the discretion of the physicians.

Main objective: To verify the value of ILR in assessing the mechanism of syncope and the efficacy of the ILR-guided therapy after syncope recurrence.

Secondary objectives:

1. To define the exact mechanism of syncope in patients with suspected or certain neurally-mediated syncope based on the initial evaluation;
2. To prospectively evaluate the correlation between tilt-induced syncope, ATP-induced asystolic response and/or carotid sinus hypersensitivity and ILR-documented spontaneous syncope associated with bradycardia and/or asystole;
3. To assess the relationship between asymptomatic and symptomatic asystoles;
4. To assess the effectiveness of pacing therapy for preventing syncope recurrence in patients implanted with a pacemaker after an ILR-documented syncope associated with asystole/bradycardia.

Inclusion criteria:

* Suspected or certain neurally-mediated syncope, based on the Guidelines of the ESC TF on Syncope.
* 3 syncope episodes in the last 2 years.
* Severe clinical presentation of syncope requiring treatment initiation in the judgement of the investigator.
* Age >30 years.
* Patients have undergone carotid sinus massage, and ILR implantation.

Exclusion criteria:

* ILR not implanted for any reason; in this case, the patients are still followed in the ILR-not implanted group.
* Carotid sinus syndrome.
* Suspected or certain cardiac syncope.
* Symptomatic orthostatic hypotension diagnosed by standing blood pressure measurement.
* Loss of consciousness different from syncope (e.g. epilepsy, psychiatric, metabolic, drop-attack, TIA, intoxication, cataplexy).
* Steal syndrome.
* Psychologically or physically (due to any other illness) unfit for participation in the study according to the opinion of the investigator.
* Patient compliance doubtful.
* Patients who are geographically or otherwise inaccessible for follow-up.
* Patient unwilling or unable to give informed consent;
* Pregnancy.
* Life expectancy < 1 year due to non-cardiac cause.

Primary endpoints: Phase 1: first ECG-documented syncope Phase 2: first syncope recurrence after implementation of ILR-guided therapy

Secondary endpoints: Phase 1:

* Asymptomatic ILR-documented arrhythmia
* ILR-documented pre-syncope/s

Phase 2:

* Total number of syncopal recurrences
* Pre-syncope recurrence

Study duration: ISSUE 2 will enroll a minimum of 400 patients during an anticipated period of 3 years. As the study will continue for a period of 6 months after the enrollment of the last patient, total study duration will be approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or certain neurally-mediated syncope, based on the Guidelines of the ESC TF on Syncope.
* 3 syncope episodes in the last 2 years.
* Severe clinical presentation of syncope requiring treatment initiation in the judgement of the investigator.
* Age >30 years.
* Patients have undergone carotid sinus massage, and ILR implantation.

Exclusion Criteria:

* ILR not implanted for any reason; in this case, the patients are still followed in the ILR-not implanted group.
* Carotid sinus syndrome.
* Suspected or certain cardiac syncope.
* Symptomatic orthostatic hypotension diagnosed by standing blood pressure measurement.
* Loss of consciousness different from syncope (e.g. epilepsy, psychiatric, metabolic, drop-attack, TIA, intoxication, cataplexy).
* Steal syndrome.
* Psychologically or physically (due to any other illness) unfit for participation in the study according to the opinion of the investigator.
* Patient compliance doubtful.
* Patients who are geographically or otherwise inaccessible for follow-up.
* Patient unwilling or unable to give informed consent;
* Pregnancy.
* Life expectancy < 1 year due to non-cardiac cause

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2002-06; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Menozzi, MD, Principal Investigator — Department of Interventional Cardiology, Opsedle S Maria Nuova, Reggio Emilia; Michele Brignole, MD, Principal Investigator — Department of Cardiology, Arrhythmologic Centre, Ospedali del Tigullio, Lavagna; Richard Sutton, MD, Principal Investigator — Royal Brompton & National Heart Hospital, London
Locations (3):
- Italy (2):
  - Department of Cardiology, Arrhythmologic Centre, Lavagna, Genova
  - Arcispedale S Maria Nuova, Reggio Emilia, Reggio Emilia
- Royal Brompton Hospital, London SW3 6NP, United Kingdom

REFERENCES:
- [Background] Steering Committee of the ISSUE 2 study. International Study on Syncope of Uncertain Etiology 2: the management of patients with suspected or certain neurally mediated syncope after the initial evaluation rationale and study design. Europace. 2003 Jul;5(3):317-21. doi: 10.1016/s1099-5129(03)00048-5. PMID 12842651
- [Result] Brignole M, Sutton R, Menozzi C, Garcia-Civera R, Moya A, Wieling W, Andresen D, Benditt DG, Vardas P; International Study on Syncope of Uncertain Etiology 2 (ISSUE 2) Group. Early application of an implantable loop recorder allows effective specific therapy in patients with recurrent suspected neurally mediated syncope. Eur Heart J. 2006 May;27(9):1085-92. doi: 10.1093/eurheartj/ehi842. Epub 2006 Mar 28. PMID 16569653